CLINICAL TRIAL: NCT07088562
Title: Evaluation of the Effectiveness of Ultrasonography-Guided Pulsed Radiofrequency to the Suprascapular Nerve in the Treatment of Adhesive Capsulitis in Elderly Patients
Acronym: pain
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Altun, pain specialist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: Radiofrequency, shoulder pain
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Capsulitis, Adhesive; Pulsed Radiofrequency; Eldery People; Ultrasound Guided Injection
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Evaluation of the Effectiveness of Ultrasonography-Guided Pulsed Radiofrequency to the Suprascapular

SUMMARY:
Adhesive Capsulitis (AC) is a condition that restricts the passive and active range of motion of the shoulder joint, impairing quality of life and activities. AC, which can be progressive and last a long time, is also called "frozen shoulder." The incidence of AC is 2-4% in the normal patient population. This rate varies between 10-30% in diabetic patients. The limitation and pain in AC joint range of motion (ROM) can last up to 3 years. There is no clear data on its prevalence in elderly patients. Its etiopathogenesis has not been fully elucidated. Fibrotic contractures form in the joint capsule. Diabetes, female gender, autoimmune diseases, thyroid disorders, immobilization, cardiovascular and cerebrovascular diseases, and advanced age are among the risk factors . AC is often diagnosed by physical examination and exclusion of other joint pathologies. Magnetic resonance imaging (MRI) can be helpful in diagnosis .

Physical therapy, medical, interventional methods, and surgery are used in the treatment of AC. In physical therapy, exercises and modalities aimed at increasing ROM are used, while medical treatment includes oral analgesics, myorelaxants, and topical analgesics. Effective treatment options include intra-articular steroid injections and radiofrequency applications for blocking the suprascapular nerve (SN). The SN originates from the ventral branches of the C5-C6 brachial plexus. It is responsible for 70% of the shoulder innervation, particularly to the shoulder joint and capsule, and the acromioclavicular joint (ACJ). It provides motor innervation to the supraspinatus and infraspinatus muscles. NS block or radiofrequency applications are frequently used in the treatment of pain in shoulder joint pathologies, impingement syndrome, and ACJ pathologies. Previously, conventional radiofrequency applied at high temperatures had destructive effects on the nerve. While conventional methods are currently used in some cases, pulsed radiofrequency is effectively applied at lower temperatures, particularly to prevent motor damage .

In this study, we aimed to present the effectiveness of pulsed radiofrequency (SS-PRF) application to the suprascapular nerve in a difficult and challenging patient group (elderly patients) in AC, a difficult disease to treat.

DETAILED DESCRIPTION:
Patients over the age of 65 who met the diagnostic criteria for AC based on clinical, radiological (MRI), and physical examination between June 2022 and June 2023, but who failed to achieve adequate pain palliation despite appropriate medical and physical therapy modalities, and who underwent SS-PRF treatment will be retrospectively reviewed. Data from the patient files will be recorded for age, gender, body mass index (BMI), symptom duration, affected side, and the presence of concomitant diabetes. Procedure: Under appropriate monitoring conditions, patients who benefited >50% from the diagnostic block received a single session of SS-PRF at 420°C (45 V, 20 ms) for 240 seconds in a semi-sitting position under ultrasound guidance after obtaining responses from the suprascapular notch with a 100 mm-long, 10 mm active-tip radiofrequency needle.

Patients whose data can be accessed through their files will have their age, gender, body mass index (BMI), symptom duration, painful side, and medical treatments recorded. Activity and Rest Numerical Rating Scale (NRS-11) and Shoulder Pain and Disability Index (SPADI) scores will be recorded before and after treatment, at weeks 4 and 12.

The NRS-11 is an 11-point numerical scale that allows patients to rate their pain from 0 (no pain) to 10 (the most severe pain they have ever experienced).

The SPADI is a validated index consisting of 13 questions, 5 assessing pain and 8 assessing disability, and scored from 0 to 100 to assess shoulder pain and functionality. Higher scores indicate greater pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 65 who were diagnosed with adhesive capsulitis through clinical physical examination and imaging and who underwent shoulder SS-PRF.
* Patients with complete data to be scanned in their files.

Exclusion Criteria:

Patients with a history of shoulder surgery,

* shoulder impingement syndrome, osteoarthritis, or other primary shoulder pathologies that could explain shoulder pain,
* patients who received shoulder injections within the last 3 months,
* patients with psychosis,
* patients with pacemakers (ICDs), patients with decompensated chronic diseases,
* patients with bleeding disorders,
* patients with active malignancy or infection,
* patients with advanced cervical disc herniation,
* patients with allergies to the medications to be administered,
* patients who could not be communicated with, and patients who did not accept the procedure were excluded from the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over the age of 65 who met the AK diagnostic criteria through clinical, radiological (MRI) and physical examination between June 2022 and June 2023, and who received SS-PRF treatment and who could not achieve adequate pain palliation despite medical and physical therapy modalities within an appropriate period of time, will be retrospectively screened.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
numerical rating scale (NRS-11) | 12 weeks
  The NRS-11 is an 11-point numerical scale on which patients can rate their pain from 0 (no pain at all) to 10 (the most severe pain they have ever felt).
shoulder pain and disability index (SPADI) | 12 weeks
  The SPADI is a validated index consisting of 13 questions, 5 of which assess pain and 8 assess disability, and is scored from 0 to 100 to assess shoulder pain and functionality. As the score increases, pain and disability increase.

CONTACTS AND LOCATIONS:
Overall Officials: halil ibrahim altun, Principal Investigator — Kanuni Sultan Süleyman Training and Research Hospital
Locations (1):
- İKanuni Sultan Süleyman Training and Research Hospital, Küçükçekmece, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided